CLINICAL TRIAL: NCT07239856
Title: Digestive Tolerance and Nutrient Absorption Kinetics of Goat Milk Versus Cow Milk in Individuals With Reported Cow's Milk Intolerance : a Controlled Single-blinded Crossover Trial
Brief Title: Goat vs. Cow Milk Digestive Tolerance
Acronym: DIGIGOAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: DIGIGOAT
Record Dates: First submitted 2025-09-11; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-05

CONDITIONS: Milk Intolerance; Milk Hypersensitivity; Cow Milk Protein Sensitivity
Keywords: Digestive confort; Goat milk; Cow milk; Stable isotopes; Milk hypersensitivity; Milk intolerance; Digestion
MeSH Terms: conditions — Lactose Intolerance; Milk Hypersensitivity | interventions — Milk

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cow milk intolerant (Experimental): Individuals who report being intolerant to cow's milk but not to goat's milk
  Interventions: Other: Cow milk; Other: Goat Milk
- Control (Experimental): Individuals who report being tolerant to both cow's milk and goat's milk.
  Interventions: Other: Cow milk; Other: Goat Milk

INTERVENTIONS:
Other: Cow milk — Consuption of 500 ml of aromatized cow milk, labeled with stable isotopes: nitrogen-15 and deuterium. Body composition is measured via bioelectrical impedance. A venous catheter is inserted. Blood, urine and breath samples are taken pre-meal, and regularly during 8 hours. Digestive tolerance and hunger are assessed using questionnaires.
Other: Goat Milk — Consuption of 500 ml of aromatized goat milk, labeled with stable isotopes: nitrogen-15 and deuterium. Body composition is measured via bioelectrical impedance. A venous catheter is inserted. Blood, urine and breath samples are taken pre-meal, and regularly during 8 hours. Digestive tolerance and hunger are assessed using questionnaires.

SUMMARY:
The objective of this study is to assess to what extent goat's milk is better tolerated than cow's milk among individuals who report being intolerant to cow's milk, and, if so, to understand the underlying factors. To achieve this, digestive discomfort sensations and postprandial kinetics of nutrients after ingestion of cow's or goat's milk will be compared in two populations: individuals intolerant to cow's milk but not to goat's milk, and individuals who show no symptoms of intolerance to either cow's or goat's milk. For this purpose, approaches based on stable isotope labeling of milk will be employed.

DETAILED DESCRIPTION:
Objective:

Although milk has many nutritional benefits, such as being rich in high-quality proteins and calcium, some people limit or exclude its consumption due to poor digestive tolerance. Lactose intolerance is a well-known cause, but other factors may occur, remaining poorly understood. Goat milk is perceived by consumers as causing fewer intestinal issues than cow milk, particularly for sensitive individuals. However, there is little scientific evidence to support this perception and to confirm the supposed health benefits of goat's milk over cow's milk. The objective of this study is to assess to what extent goat's milk is better tolerated than cow's milk among individuals who report being intolerant to cow's milk, and, if so, to understand the underlying factors.

Design:

This study is crossover study, randomized for the order of testing (goat milk or cow milk), conducted in a single-blind design (participants are not informed about the test meal, which is masked by aroma), involving two groups of at least ten volunteers: individuals intolerant to cow's milk but not to goat's milk, and individuals who show no symptoms of intolerance to either cow's or goat's milk. Each subject will have consumed both milks at the end of the two sessions, with a minimum one-month interval.

Postprandial Test Procedure:

Two days before the test, subjects must exclude consumption of the main dairy products (yogurt, cheese, milk, and custard creams). Volunteers arrive in a fasted state on the investigation day and are hospitalized for one day per session. On the first visit, volunteers bring a stool sample. Upon arrival, body composition is measured via bioelectrical impedance and a venous catheter is inserted. Blood samples are taken 30 minutes pre-meal, every 30 minutes for the first 4 hours, and hourly thereafter, totaling 291 mL. Urine is collected before the meal and every 2 hours post-meal. Respiratory is measured hourly using an indirect calorimeter. Digestive tolerance and hunger are assessed hourly using questionnaires. Volunteers remain semi-reclined for about 9 hours and fast until the experiment ends, receiving hourly water.

The test meal consists of aromatized 500 ml of cow's or goat's milk, labeled with stable isotopes: nitrogen-15 and deuterium. The incorporation rate is minimal and safe for human health, commonly used in clinical studies. The 15N enrichment is measured in collected biological samples (blood, urine) to track the digestive and metabolic fate of dietary amino acids, enabling precise evaluation of nutrient availability kinetics in the body. After the investigation day, volunteers can go home post-meal. A follow-up call the next day checks for digestive symptoms, with the doctor assessing the need for symptomatic treatment.

The protocol has been approved by the Ethical Committee and authorized by the French Agency of Drugs and Health. The personal data management will be in accordance with the regulation on personal data protection ("regulation n° 2018-493 du 20 juin 2018").

ELIGIBILITY:
Inclusion Criteria:

* Individuals who report being intolerant to cow milk but not to goat milk (one group) or tolerant to both cow milk and goat milk (another group)
* Good general health (WHO grade = 0)
* Affiliated with a social security scheme
* Free, informed, and express consent, in accordance with the public health code: 'No research mentioned in 2° of Article L. 1121-1 can be conducted on a person without their free, informed, and express consent.

Exclusion Criteria:

* Individuals under guardianship or curatorship
* Individuals under legal protection
* Any known food allergies
* Anemia: hemoglobin levels below 13 g/dL for men and 12 g/dL for women
* Pregnant women or those likely to be (based on a positive urine pregnancy test at the time of inclusion)
* Excessive alcohol consumption (>2 drinks/day). Harmful alcohol consumption is assessed by the investigator at the time of inclusion.
* Hypertension, diabetes, digestive tract diseases (except for irritable bowel syndrome, IBS), liver or kidney diseases, severe heart disease. The presence of these conditions will be assessed by the investigator based on usual clinical criteria and the volunteers' declarations during inclusion. Hypertension: Significant arterial hypertension as determined by the investigator or systolic blood pressure greater than or equal to 140 mmHg and/or diastolic blood pressure greater than or equal to 90 mmHg on the day of inclusion. Diabetes: Type 1 or Type 2 diabetes or any fasting blood glucose level > 1.25 g/l. Digestive tract disease: Gastrointestinal disorders deemed by the investigator as clinically significant (bleeding, vomiting, constipation/diarrhea grade >1), any inflammatory bowel disease, acute gastroenteritis in the month preceding the intervention. Liver disease: Any significant liver disorder as determined by the investigator or any AST/ALT > 2.5 times the upper normal limit.
* Elite athletes (> 8 hours per week)
* Blood donation in the 3 months preceding the start of the study
* Participation in a clinical study in the 3 months preceding the study
* Lack of free, informed, and express consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Digestive discomfort score from 0 to 8 hours post-meal | 0, 1, 2, 3, 4, 5, 6, 7, 8 hours post-meal
  A digestive tolerance questionnaire (Casellas, 2009) and a hunger sensation questionnaire using visual analog scales are administered hourly. These are based on scales from 1 to 10 to assess feelings of : flatulence, nausea, diarrhea, bloating, and abdominal pain.

SECONDARY OUTCOMES:
15N enrichment of plasma and urine fractions from 0 to 8 hours post-meal | 0, 1, 2, 3, 4, 5, 6, 7, 8 hours post-meal
  The measurement of isotopic enrichment of nitrogenous compounds in plasma and urine, in response to the ingestion of 15N-labeled milk proteins, provides an estimate of proteins absorption kinetic.
2H enrichment of plasma fatty acids from 0 to 8 hours post-meal | 0, 1, 2, 3, 4, 5, 6, 7, 8 hours post-meal
  The measurement of isotopic enrichment of fatty acids in plasma, in response to the ingestion of 2H-labeled milk lipids, provides an estimate of fatty acid absorption kinetics.
2H enrichment of plasma glucose from 0 to 8 hours post-meal | 0, 1, 2, 3, 4, 5, 6, 7, 8 hours post-meal
  The measurement of isotopic enrichment of glucose in plasma, in response to the ingestion of 2H-labeled milk lactose, provides an estimate of lactose absorption kinetics.
Blood metabolites concentrations from 0 to 8 hours post-meal | 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 7, 8 hours post-meal
  Analysis of the amino acid, urea, glucose, triglyceride, free fatty acid, cholesterol, and insulin concentrations in blood
Exhaled breath gas concentrations from 0 to 8 hours post-meal | 0, 1, 2, 3, 4, 5, 6, 7, 8 hours post-meal
  Hydrogen (H2), methane (CH4), and carbon dioxide (CO2) concentration from exhaled air
Substrate oxidation rates from 0 to 8 hours post-meal | 0, 1, 2, 3, 4, 5, 6, 7, 8 hours post-meal
  Fat and glucose oxidation are assessed by measuring respiratory exchanges using indirect calorimetry
Intestinal microbiota composition | Once at the beginning of enrollement
  Volunteers must bring a stool sample in the container previously provided to them. The samples will be analyzed using the 16S rRNA method to assess gamma and beta diversity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Avicenne, 125 rue de Stalingrad, Bobigny, France

IPD SHARING:
Plan to Share IPD: No